CLINICAL TRIAL: NCT02288975
Title: The Effect of Early Cytokine Absorption on the Systemic Inflammatory Response Syndrome and Organ Dysfunction in the First 48 Hours of Septic Shock
Brief Title: Adsorbtion of Cytokines Early in Septic Shock: the ACESS Study
Status: Completed | Type: Observational
Sponsor: Zsolt Molnár, MD, PhD, DEAA (Other)
Responsible Party: Sponsor-Investigator, Zsolt Molnár, MD, PhD, DEAA, Ph.D. student; Department of Anaesthesiology and Intensive Therapy, Szeged University
Organization: Szeged University (Other)
Other Study IDs: CytoSorb-2014
Record Dates: First submitted 2014-11-05; First posted 2014-11-13 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Sepsis; Septic Shock
Keywords: hemoadsorption; extracorporeal blood purification; CytoSorb; hemofiltration; SIRS; sepsis; septic shock; membranes; ICU; dialysis; adsorption
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CytoSorb: Patients with septic shock will get routine ICU care supported by CytoSorb® treatment.
  Interventions: Device: CytoSorb 300ml device (3804606CE01)
- Control: Patients with septic shock will get routine ICU care.

INTERVENTIONS:
Device: CytoSorb 300ml device (3804606CE01)
  Groups: CytoSorb

SUMMARY:
The aim of the study is to investigate the effect of CytoSorb® treatment within the first 48 hours of septic shock on organ dysfunction, microcirculation and on the cytokine storm as monitored by leukocyte activation and inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

* Signs of hypoperfusion: serum lactate >2 mmol/L, low central venous oxygen saturation (ScvO2) (<70%) or high ScvO2 (>85%), metabolic acidosis, oligo-anuria, high venous-to-arterial CO2-gap (dCO2 >6 mm Hg)
* Hemodynamic support with vasopressors
* Procalcitonin level ≥ 3 ng/ml
* Invasive hemodynamic monitoring
* Written informed content

Exclusion Criteria:

* Patients under 18 years
* Pregnancy (bHCG test positivity)
* Surgical intervention in context with the septic insult
* New York Heart Association IV heart failure
* Acute coronary syndrome
* Need for acute or chronic hemodialysis
* Acute haematological malignancies
* Cardiogenic shock
* Post cardiopulmonary resuscitation care
* Immunosuppression, systemic steroid therapy (>10mg prednisolon/day)
* Human immunodeficiency virus infection (HIV) and active AIDS
* Patients with donated organs
* Thrombocytopenia (<20.000/ml)
* More than 10%-of body surface area with third degree burn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with septic shock of medical origin
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cytokine response | First 48 hours of septic shock
  Cytokine response: procalcitonin, C-reactive protein, interleukin-1, interleukin-1ra, interleukin-6, interleukin-8, interleukin-10, Tumor Necrosis Factor- α
Organ dysfunctions | First 48 hours of septic shock
  Organ dysfunctions: SOFA-scores, neurologic function (Glasgow coma scale), hemodynamic function (PiCCO parameters, ScvO2, lactate, dCO2), pulmonary function (gas exchange, pulmonary mechanics, Acute Respiratory Distress Syndrome classification (BERLIN)), renal function (KDIGO-, RIFLE-scores), gastrointestinal function (liver, GIT function, hematology (hemostasis, qualitative blood count)

SECONDARY OUTCOMES:
Leukocyte function | First 48 hours of septic shock
  Leukocyte function: heterogeneity of leukocyte cell population in the bloodstream, T-cell activation and apoptosis, leukocyte inflammatory markers expression
Microcirculation | First 48 hours of septic shock
  Microcirculation: orthogonal polarization spectroscopy (OPS), gastric tonometry

OTHER OUTCOMES:
Length of intensive care unit stay, | First 48 hours of septic shock
Length of hospital stay | First 48 hours of septic shock
Mortality | First 48 hours of septic shock

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Intensive Therapy, Szeged, Csongrád megye, Hungary

REFERENCES:
- [Derived] Hawchar F, Laszlo I, Oveges N, Trasy D, Ondrik Z, Molnar Z. Extracorporeal cytokine adsorption in septic shock: A proof of concept randomized, controlled pilot study. J Crit Care. 2019 Feb;49:172-178. doi: 10.1016/j.jcrc.2018.11.003. Epub 2018 Nov 10. PMID 30448517